CLINICAL TRIAL: NCT02501772
Title: The Evaluation of Effect of Sanyinjiao (SP6) Acupressure on Early Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chunag Shih-Ming, Mackay Memorial Hospital, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14MMHIS139
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sanyinjiao acupressor group (Experimental): In addition to maintain current treatment included oral anti-hyperglycemia agent and ACEI(angiotensin-converting enzyme inhibitor ) or ARB, subjects should wear ankle band at Sanyinjiao point ( calf , ankle on the foot tip 3 inch ), with the thumb pressing daily five minutes later and carry more than four hours for 8 weeks
  Interventions: Device: acupressure by ankle band
- Control Group (Sham Comparator): In the control group, ankle band was place as same as the those for the SA(Sanyinjiao acupressor) group, but was wearing at the acupoint of Sanyinjiao with anti- surface without pressure. It was applied four hours per day for 8 weeks
  Interventions: Device: acupressure by ankle band

INTERVENTIONS:
Device: acupressure by ankle band

SUMMARY:
For diabetic patient with persisted albuminuria under the intensive control on blood pressure and blood glucose, the non-invasive method of acupressure at Sanyinjiao (SP6) is easy to use and significantly effect on albuminuria reduction in patients of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 and 80 years old;
2. HbA1c was lower than 9% according to the NGSP(National Glycohaemoglobin Standardisation Programme);
3. estimated glomerular filtration rate (eGFR) was more than 60 mL/min/1.73 m2.

Exclusion Criteria:

1. Hyperglycemic crisis, including HHS(hyperglycemic hyperosmolar syndrome) and DKA(diabetic ketoacidosis );
2. Persist diabetes poorly control, Hemoglobin A1c [HbA1c] >9%;
3. Endocrine disorders: such as abnormal function of thyroid, pituitary, and sex glands;
4. heart diseases:such as arrhythmia, myocardial infarction, heart failure, or installed pacemaker;
5. immune and allergic diseases: such as systemic lupus erythematosus and asthma;
6. liver or kidney dysfunction: GOT or GPT(glutamate-pyruvate transaminase ) > 80 IU/L, eGFR<60 (mL/min);
7. pregnant or lactating women;
8. less than 6months postpartum;
9. acute illness, fever, Lower urinary tract infection, NSAID(nonsteroidal antiinflammatory drug) administration;
10. physical dysfunction because of stroke.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
urinary spot albumin creatine excretion ratio (UACR) change | 8 week duratoin

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memerial Hospital, Taipei, Taiwan